CLINICAL TRIAL: NCT06841627
Title: Exploring the Mechanism of Osteopathic Manual Therapy (OMT) on Brain Structure and Function in Primary Headache Patients: A Pilot Study
Brief Title: Osteopathic Manual Therapy (OMT) and Brain Structure and Function in Primary Headache Patients: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: Auburn University MRI Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000226; 2254326-1 (Other: Edward Via College of Osteopathic Medicine)
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Primary Headaches (Migraines, Tension, Cluster Headaches)
Keywords: Migraine; Headaches; Osteopathic Manipulative Treatment; Brain; OMT
MeSH Terms: conditions — Migraine Disorders; Cluster Headache; Headache | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMT Treatment Group (Experimental)
  Interventions: Other: Osteopathic Manipulative Therapy

INTERVENTIONS:
Other: Osteopathic Manipulative Therapy — Evaluation looking for Somatic Dysfunction (SD) involving the head, neck, upper thoracic spine, rib cage and sacroiliac joint. OMT techniques will include a mix of the following: Osteopathic Cranial Manipulative Medicine, Muscle Energy Technique, Facilitated Positional Release, Indirect Myofascial Release, and Counterstrain.

SUMMARY:
Chronic headaches are associated with changes in brain structure and function that may be associated with increased suffering and disability. Understanding how Osteopathic Manipulative Therapy (OMT) affects these changes would reveal new insight into how the brain processes pain and returns to normal function. Also, demonstrating these changes would provide evidence regarding how OMT causes a reduction in pain and disability, supporting the recommendation for OMT as a primary treatment option for headaches.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of primary headache (migraine, tension-type, cluster) from a healthcare provider
* have experienced at least one headache episode a month for the previous 1 year (or longer)
* age of PH onset was less than 50 years, currently taking medication for headaches.

Exclusion Criteria:

* presence of headaches due to some other underlying medical condition (secondary headaches)
* traumatic brain injury
* fibromyalgia, epilepsy
* diagnosis of a neurodegenerative disorder
* history of brain tumor or cancer
* history of cervical radiculopathy (pinched nerve in the neck)
* currently undergoing manual therapy type treatment or have a a treatment within 2 weeks of enrollment(chiropractic, OMT, massage, PT)
* currently pregnant
* have had an injection to treat headaches within the previous 3 months from study enrollment
* contraindications to MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Brain Structural and Functional Changes | From enrollment to the end of treatment at 5 weeks
  Structural MRI will assess physical changes in brain anatomy, including differences in the size, shape, or density of specific brain regions. For example, changes in gray matter volume or white matter integrity may indicate neuroplasticity changes response to an OMT. Functional MRI (fMRI) will measure brain activity by detecting changes in blood flow within the central pain network. When a specific brain region becomes more active, it requires more oxygen, which fMRI can detect. This will help determine whether the intervention alters brain function, such as increased activation in areas involved in movement, memory, or pain processing. Magnetic Resonance Spectroscopy (MRS), unlike standard MRI, which provides images of brain structures, will analyze chemical changes in the brain. It detects levels of important brain metabolites involved in neural signaling neuronal health.

SECONDARY OUTCOMES:
Headache Impact Test - 6 (HIT-6) | From enrollment to the end of treatment at 5 weeks
  The HIT-6 (Headache Impact Test-6) measures how headaches affect daily life, including pain severity, frequency, and impact on work and social activities.
Short Form -36 (SF-36) | From enrollment to the end of treatment at 5 weeks
  The SF-36 (Short Form-36 Health Survey) is a 36 question survey that assesses overall physical and mental well-being, evaluating factors like physical function, pain, energy levels, and emotional health.
Depression Anxiety and Stress Scale 21 (DASS-21) | From enrollment to the end of treatment at 5 weeks
  The DASS-21 (Depression, Anxiety, and Stress Scale-21) is a 21 question survey that examines emotional well-being by measuring levels of depression, anxiety, and stress.
Headache intensity | From enrollment to the end of treatment at 5 weeks
  Headache intensity will be measured by an 11 point numerical rating scale from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cawley, DC, Principal Investigator — Edward Via College of Osteopathic Medicine
Locations (1):
- Auburn University MRI Center and Edward Via College of Medicine, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No